CLINICAL TRIAL: NCT02226510
Title: MetfoRmin and Its Effects on Myocardial Dimension and Left Ventricular Hypertrophy in Normotensive Patients With Coronary Artery Disease
Brief Title: MetfoRmin and Its Effects on Left Ventricular Hypertrophy in Normotensive Patients With Coronary Artery Disease
Acronym: MET-REMODEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013CV08; 2014-003189-26 (EudraCT Number); 14/ES/1061 (Other: REC)
Record Dates: First submitted 2014-08-18; First posted 2014-08-27 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Left Ventricular Hypertrophy; Insulin Resistance; Coronary Artery Disease; PreDiabetes
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Insulin Resistance; Coronary Artery Disease; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules (with an identical appearance to the active drug) and containing only microcrystalline cellulose PhEur
  Interventions: Drug: Placebo
- Metformin XL (Active Comparator): In the active arm, the added therapy will be metformin XL in an initial dose of 1000mg/day (metformin XL 500mg x2/day). They will continue on Metformin XL 500mg x2/day for two weeks and after safety blood checks the metformin XL dose will be increased to 2000 mg/day. If the higher dose cannot be tolerated the dose will be reduced to 1000mg/day (and stopped if this cannot be tolerated).
  Interventions: Drug: Metformin XL

INTERVENTIONS:
Drug: Metformin XL — In the active arm, the added therapy will be metformin XL in an initial dose of 1000mg/day . They will continue on Metformin XL 500mg x2/day for 2 weeks and after safety blood checks the metformin XL dose will be increased to 2000 mg/day. If the higher dose cannot be tolerated the dose will be reduced to 1000mg/day.
  Other Names: Diagemet XL
  Arms: Metformin XL
Drug: Placebo — Placebo capsules (with an identical appearance to the active drug) containing only microcrystalline cellulose PhEur will be administered.
  Arms: Placebo

SUMMARY:
Thickening of the heart muscle (left ventricle) known medically as Left Ventricular Hypertrophy (LVH) is very common in patients with heart disease. This increases risk of cerebrovascular/cardiovascular event.

LVH is asymptomatic and managed by the use of medication to control blood pressure, however LVH may be seen in normotensive patients where factors such as obesity and insulin resistance are present.

Insulin resistance is a condition where although the body produces insulin it is unable to utilize it effectively. Metformin, a drug used to treat diabetes, can reduce insulin resistance and cause weight loss, it may therefore improve LVH. This study will investigate the ability of metformin to reduce LVH in patients with heart disease, this may be a novel way forward in the risk reduction of cerebrovascular/cardiovascular events. Participants will be identified throughout NHS Tayside, those eligible will be randomly allocated to either metformin or a dummy medication (placebo) and will receive one year of treatment. At the beginning of the study, the thickness of the heart muscle will be measured by ultrasound scan and cardiac Magnetic Resonance Imaging (cMRI). We will also perform non-invasive tests to measure blood vessel function. These tests will be repeated after one year. At the end of the study, we will investigate the difference between placebo treatment and metformin treatment.

This study is funded by the British Heart Foundation.

DETAILED DESCRIPTION:
This is a single centre trial designed to investigate the benefit, if any, of 12 month metformin XL 2000mg/day treatment on left ventricular hypertrophy (LVH) in 64 nondiabetic participants with Ischaemic heart disease (IHD) and insulin resistance (IR) and/or prediabetes.

Participants will be seen on seven occasions: screening, baseline/randomisation, 2 weeks post randomisation, month 1, month 4, month 8 and final month 12, during which vital signs and safety bloods will be performed. There will also be three telephone visits at: month 2, month 6 and month 10.

At a screening visit an initial history will be performed following informed consent. Participants will then undergo an echocardiogram (a painless ultrasound scan of the heart) in the Department of Clinical Pharmacology, Ninewells Hospital, Dundee. Blood pressure will be recorded and blood tests to determine fasting insulin resistance index (FIRI), prediabetes and routine safety, prior to metformin administration, will be performed.

Participants who meet all inclusion criteria will return for the randomisation visit within 4 weeks of screening where a Cardiac Magnetic Resonance Imaging (cMRI) scan will be performed followed by randomisation to either Metformin XL or placebo in a double blind, randomised fashion. Also, at this visit endothelial function tests will be performed to assess peripheral blood vessels in the forearm, central obesity will be quantified using waist circumference and waist to hip ratio (WHR) and study specific blood sampling performed (with participant consent).

At the final visit or early withdrawal the following will be performed: vital signs, safety bloods, study specific bloods (with participant consent), echocardiography, endothelial function tests and cMRI.

In the active arm, therapy will be metformin XL in an initial dose of 1000mg/day (metformin XL 500mg x2/day). Participants will continue on Metformin XL 500mg x2/day for two weeks, following safety blood checks this dose will be increased to 2000 mg/day. If the higher dose cannot be tolerated it will be reduced to 1000mg/day (or stopped if not tolerated).

The target dose of metformin XL at 2000mg/day was chosen based on a previous study of metformin in nondiabetic heart failure patients with IR, this study demonstrated a beneficial effect of metformin on insulin resistance, weight reduction and an improvement in submaximal exercise. The study used the immediate release form of metformin (target of 1000 mg x2/day) which was associated with significant gastrointestinal side effects resulting in 13% withdrawal of study medication. For this reason we have selected metformin XR due to improved gastrointestinal tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Participant willing and able to give informed consent.
* Documented Ischaemic Heart Disease: either angio-graphically documented coronary artery disease or a previous history of myocardial infarction/angina.
* Screening echocardiography based diagnosis of LVH (LV mass indexed to height to the allometric power of 1.7; males > 81g/h1.7, females >60g/h1.7)
* Fasting insulin resistance index ≥ 2.7 AND/OR HbA1c >5.6 and less than 6.5 at screening
* Blood pressure < 140/85 mm Hg or 24hr BP <135/85 daytime average in screening
* Able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Cognitive impairment
* Type 1 or 2 Diabetes mellitus
* Chronic Heart Failure as evidenced by echocardiogram or documented diagnosis of CHF
* Left Ventricular Ejection Fraction <45% on screening echocardiography
* Contraindications to cardiac MRI (pacemakers, claustrophobia, metal implants, history of penetrative eye injury or exposure to metal fragments in eye requiring medical attention)
* Malignancy (receiving active treatment) or other life threatening disease, renal disease (CKD class 3B or worse)
* Pregnancy/lactating females
* Any other reason considered inappropriate by a study physician
* Participants who have participated in any other clinical trial within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Mass Index | 12 months
  Cardiac magnetic resonance imaging will be performed at baseline and at 12 months, to measure Left Ventricular Mass Index in patients

SECONDARY OUTCOMES:
Central and Abdominal obesity | 12 months
  Abdominal magnetic resonance imaging will be performed at baseline and at 12 months to measure the changes in central and abdominal obesity
Left Ventricular end systolic volume, | 12 months
  Cardiac magnetic resonance imaging will be performed at baseline and at 12 months to measure Left Ventricular end systolic volume
Endothelial Function | 12 months
  Improvement in endothelial function with metformin compared with placebo, measured by FMD and PWA and skin reactive hyperaemia
Insulin Resistance / Prediabetes | 12 months
  Improvement in insulin resistance (IR)/ prediabetes when treated with metformin compared to placebo in patients with IHD and IR measure using Fasting Insulin Resistance Index (FIRI)
Inflammatory and other cardiovascular blood markers | 12 months
  Changes in inflammatory and other cardiovascular blood markers such as BNP/F2 Isoprostanes/oxi-LDL/Troponin T, when treated with metformin compared to placebo in patients with IHD and IR
Number of participants with Adverse Event | 12 months
  Safety and efficacy of Metformin XL will be determined by monitoring changes from randomisation till the end of the study or so long the patient remains in the study, whichever is earlier.
Left Ventricularend diastolic volume | 12 months
  Cardiac magnetic resonance imaging will be performed at baseline and at 12 months to measure Left Ventricular end diastolic volume
Left Ventricular Ejection Fraction | 12 months
  Cardiac magnetic resonance imaging will be performed at baseline and at 12 months to measure Left Ventricular Ejection Fraction
Left Ventricular Mass | 12 months
  Cardiac magnetic resonance imaging will be performed at baseline and at 12 months to measure Left Ventricular Mass

CONTACTS AND LOCATIONS:
Overall Officials: Chim Lang, MD, Principal Investigator — University of Dundee
Locations (1):
- Ninewells Hospital & Medical School, Dundee, Angus, United Kingdom

REFERENCES:
- [Derived] Mohan M, McSwiggan S, Baig F, Rutherford L, Lang CC. Metformin and its effects on myocardial dimension and left ventricular hypertrophy in normotensive patients with coronary heart disease (the MET-REMODEL study): rationale and design of the MET-REMODEL study. Cardiovasc Ther. 2015 Feb;33(1):1-8. doi: 10.1111/1755-5922.12101. PMID 25545400

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT02226510/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT02226510/SAP_001.pdf